CLINICAL TRIAL: NCT01384838
Title: Randomized Trial of Exercise Training in Postmenopausal Patients With Hormone-receptor Positive Breast Cancer Undergoing Treatment With Aromatase Inhibitors
Brief Title: Exercise Training in Postmenopausal Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Daniela Wolkersdorfer, Arbeitsgemeinschaft medikamentoese Tumortherapie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AGMT_BC_Sports
Record Dates: First submitted 2011-06-28; First posted 2011-06-29 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Physical Activity
Keywords: breast cancer; physical activity; sports; exercise
MeSH Terms: conditions — Motor Activity; Breast Neoplasms | interventions — Counseling; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling (Other): Patients are to receive identical counseling for ideal nutritional, lifestyle, physical activity.
  Interventions: Behavioral: Counseling
- Controlled physical activity (Experimental): All patients are to receive identical counseling for ideal nutritional, lifestyle, physical activity.
  Patients randomized to Arm 2 will additionally undergo a controlled and observed program of physical activity for a period of 6 months. Thereafter the patients are expected to adhere to a comparable, unobserved exercise program at home.
  Interventions: Behavioral: physical activity

INTERVENTIONS:
Behavioral: Counseling — Nutritional, lifestyle and sports counseling
  Arms: Counseling
Behavioral: physical activity — counseling and controlled physical activity
  Arms: Controlled physical activity

SUMMARY:
This randomized trial aims to assess if a well defined subgroup of breast cancer patients benefit from a controlled physical activity program.

All patients will be screened for their physical ability to complete the interventional exercise program. Only patients capable and willing to take part in this study and meeting all inclusion and exclusion criteria will be randomized.

All patients are to receive identical counseling for ideal nutritional, life-style and physical activity.

Patients randomized to Arm 2 will additionally undergo a controlled and observed program of physical activity for a period of 6 months. Thereafter the patients are expected to adhere to a comparable, unobserved exercise program at home.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Postmenopausal women with hormone receptor positive breast cancer (as defined by HR >= ++ and/or PR >= ++) who are treated with aromatase inhibitors
* ECOG performance status <= 2
* all age groups

Exclusion Criteria:

* Pathologic ergometry
* Uncontrolled diabetes mellitus
* Uncontrolled hypertension
* COPD > II
* Active opportunistic infection
* NYHA heart failure III or IV

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Individual maximum power output in watt (Pmax) on a bicycle ergometer after 6 months of controlled or unobserved physical activity. | after 6 months

SECONDARY OUTCOMES:
Determination of feasibility of achieving 12 MET/week (metabolic units) on an outpatient basis | after 6 and 12 months
Evaluation of the influence of controlled/observed physical activity versus lifestyle counseling only on Fitness level, Quality of Life, rate of infections, weight, body mass index BMI, Body fat percentage | after 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, Prof.Dr., Study Director — Arbeitsgemeinschaft medikamentoese Tumortherapie
Locations (1):
- Universitätsklinik für Innere Medizin III mit Hämatologie, internistischer Onkologie, Infektologie, Rheumatologie und Onkologisches Zentrum, Salzburg, Austria

REFERENCES:
- [Derived] Westphal T, Rinnerthaler G, Gampenrieder SP, Niebauer J, Thaler J, Pfob M, Fuchs D, Riedmann M, Mayr B, Reich B, Melchardt T, Mlineritsch B, Pleyer L, Greil R. Supervised versus autonomous exercise training in breast cancer patients: A multicenter randomized clinical trial. Cancer Med. 2018 Dec;7(12):5962-5972. doi: 10.1002/cam4.1851. Epub 2018 Nov 10. PMID 30415507